CLINICAL TRIAL: NCT06665867
Title: VICO-trial: Video Consultations in the Follow-up of Children With Functional Abdominal Pain Disorders
Acronym: VICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Merit Monique Tabbers, Dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024.0101
Record Dates: First submitted 2024-07-19; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Functional Abdominal Pain Disorders; Irritable Bowel Syndrome (IBS); Functional Dyspepsia; Abdominal Migraine
Keywords: E-health; Video consultations; Children; Functional abdominal pain disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video consultation (Experimental): These participants are randomized for video consultations. Participants will receive two follow-up consultations via video.
  Interventions: Other: Video consultation
- Face-to-face consultation (Active Comparator): These participants are randomized for face-to-face consultations. Participants will receive two follow-up face-to-face consultations in the hospital.
  Interventions: Other: Face-to-face consultation

INTERVENTIONS:
Other: Video consultation — Participants will have their follow-up consultation with the physician via video. The consultation takes place via the participant's/parent's own device.
  Arms: Video consultation
Other: Face-to-face consultation — The follow-up consultation with the physician will take place at the hospital.
  Arms: Face-to-face consultation

SUMMARY:
The goal of this non-inferiority randomized controlled multi-center trial is to investigate the use of video consultations in the follow-up care of children aged 4 - 18 years old with functional abdominal pain disorders (FAPDs). Video consultations will be compared to face-to-face consultations. Clinical outcomes and patients' and parents' healthcare experience will be compared between both groups.

Primary outcome is adequate relief after 12 weeks: the hypothesis is that video consultations are not inferior to face-to-face consultations regarding clinical outcomes and that adequate relief will be the same for both groups.

Participants and/or parents will be asked to complete a diary for 1 week and a questionnaire after every consultation: at baseline, after 6 weeks and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 years to 17 years
* Meeting the Rome IV criteria for one of the four types of Functional Abdominal Pain Disorders (FAPD's): functional dyspepsia, irritable bowel syndrome, abdominal migraine, functional abdominal pain - not otherwise specified.
* Being able to conduct a video consultation

Exclusion Criteria:

* If no follow-up consultation is indicated
* If it is necessary that the follow-up consultations are face to face

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Adequate relief | After 12 weeks
  Proportion of participants reporting adequate relief. Adequate relief is a patient-reported outcome. Participants will be asked at 6 weeks and 12 weeks whether they have adequate relief of their Functional Abdominal Pain Disorder related complaints using a binary outcome (yes/no). Participants will complete a diary for a week and participants will be asked about adequate relief in the diary on day 7.

SECONDARY OUTCOMES:
Pain intensity | 12 weeks
  Number of children with a decrease of 30% of pain intensity after 12 weeks compared to baseline, measured on a Visual Analogue Scale (VAS) of 0-10. A score of 0 means no pain and a score of 10 means a lot of pain. The VAS-score is a mean score of 7 consecutive days. Children will be asked to fill in a diary for 7 days at baseline, after 6 weeks and after 12 weeks.
Pain frequency | 12 weeks
  Number of children with a decrease of 30% pain frequency per day after 12 weeks compared to baseline. Pain frequency will be recorded as number of hours of pain per day, as a mean of 7 consecutive days. Children will be asked to fill a diary for 7 days at baseline, after 6 weeks and after 12 weeks.
Healthcare experience | 12 weeks
  Both parents/guardians and children (if > 8 years old) will be asked to complete the Patient Reported Experience Measure for Specialist Medical Care questionnaire after every consultation. The questionnaire consists of 7 questions that participants can answer using a 10-point Likert scale, where a score of 1 means 'No, not at all' and a score of 10 means 'Yes, completely'. The questionnaire also contains one question with a binary answer (yes/no).
Shared decision making (parents/guardians) | 12 weeks
  Parents/guardians will be asked to complete the CollaboRATE questionnaire after every consultation. The questionnaire consists of three questions regarding shared decision making tasks during consultation. Responses to each question range from 0 ("no effort was made") to 9 ("every effort was made").
Shared decision making (children) | 12 weeks
  Children (if > 8 years old) will be asked to fill in the CollaboRATE questionnaire after every consultation. The questionnaire consists of three questions regarding shared decision making tasks during consultation. Responses to each question range from 0 ("no effort was made") to 9 ("every effort was made").
Experience of patients and parents/guardians with video consultations | 12 weeks
  Both parents/guardians and children (if > 8 years old) will be asked to fill in a questionnaire regarding their experience with the video consultation after every consultation.
Experience of healthcare professionals with video consultations | End inclusion phase (expected 1.5 years)
  Upon completion of the inclusion phase of the trial (expected 1.5 years from its start), all participating physicians will complete a questionnaire about their experience with video consultations.
Number of no shows | 12 weeks
  Proportion of no shows
Number of extra face to face consultations | 12 weeks
  Number of face to face consultations related to FAPD during the 12 week trial period, as extra to the two per protocol follow-up consultations. Participants will be asked a question in their questionnaire whether they went to the hospital (e.g. emergency department or extra consultation with their treating physician) for FAPD related complaints in the time between the two plannend consultations.
Number of hours absent from school due to consultation | 12 weeks
  Number of hours children were absent from school due to the consultation
Number of hours absent from work due to consultation | 12 weeks
  Number of work hours missed by parents/guardians due to the consultation
Duration of consultations | 12 weeks
  Duration of consultations for both face to face consultations and video consultations

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands